CLINICAL TRIAL: NCT03558984
Title: Prospective, Multicenter, Randomized, Parallel Controlled, Two Arms, Single Blind, Study to Assess the Efficacy and Safety of D-PLEX Administered Concomitantly With the SOC IV Prophylactic Antibiotic Treatment vs. SOC in Prevention of Post-Cardiac Surgery Sternal Infections
Brief Title: D-PLEX 302: Efficacy and Safety of D-PLEX in the Prevention of Sternal Infection Post Cardiac Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: company prioritization reasons
Sponsor: PolyPid Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D-PLEX 302
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Surgical Site Infection; Sternal Infection; Cardiac Surgery
Keywords: Cardiac; Surgery; Sternotomy; Heart; CABG; Valve-replacement; Aorta-replacement
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized to either the treatment arm (D-PLEX + SOC prophylactic antibiotic treatment) or to control arm (SOC prophylactic antibiotic treatment only), in a 1:1 ratio.
  Subjects will be blinded to the study arm.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded to the treatment arm assignment. The study site personnel present at the baseline procedure as well as the physician performing the procedure will be trained not to disclose the treatment arm to the subject, his/her family, to health care providers outside of the surgery department and to the study sponsor.
  Two independent of the sponsor/investigator committees will be involved in the assessment of study outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- D-PLEX + SOC (Experimental): For subjects randomized to the investigational treatment arm, D-PLEX treatment will be applied at the end of the index surgery just before closing the chest, as an adjunct to the SOC prophylactic antibiotic treatment.
  Interventions: Drug: D-PLEX; Other: Standard of Care
- Standard of Care (Other): For subjects randomized to the control arm, the surgical treatment will be as per the SOC.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: D-PLEX — D-PLEX is a new formulation of extended release of Doxycycline (active ingredient)
  Arms: D-PLEX + SOC
Other: Standard of Care — The SOC prophylactic antibiotic treatment will be consistent and standardized for all sites in the clinical study. is based on "The society of thoracic surgeons practice guideline series: antibiotic prophylaxis in cardiac surgery, part II: antibiotic choice."

SUMMARY:
Prospective, Multinational, Multicenter, Randomized, Parallel Controlled, Two arms, Single Blind, Study to Assess the Efficacy and Safety of D-PLEX Administered Concomitantly with the Standard of Care (SOC) IV Prophylactic Antibiotic Treatment vs. SOC in Prevention of Post-Cardiac Surgery Sternal Infections.

Study to assess D-PLEX efficacy and safety in preventing sternal infections over a period of 90 days (3 months) post cardiac surgery with median sternotomy, in patients with high risk for infection compared to the control arm.

DETAILED DESCRIPTION:
This is Phase III study to evaluate the anti-infective efficacy and safety of D-PLEX, a new formulation of extended release of Doxycycline, over a period of 3 months post operation by preventing sternal infection post cardiac surgery in patients above the age of 18, including high risk patients for infection. Study will be conducted in about 45 sites in US (about 15 sites), Europe and Israel, recruitment period will last about 18 months. D-PLEX will be administered as a single application. For subjects randomized to the investigational treatment arm, D-PLEX treatment will be applied at the end of the index surgery just before closing the chest, as an adjunct to the SOC prophylactic antibiotic treatment. For subjects randomized to the control arm, the surgical treatment will be as per the SOC. Pre- and post-operative care for both arms will be performed per site SOC. Patients will followed-up during 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to elective and/or urgent median sternotomy for cardiac surgery, who are preoperative hemodynamically stable.
2. Males and females.
3. Subjects age of 18 and older.
4. Subjects with both Diabetes Mellitus AND BMI≥30 OR

   Diabetes Mellitus/BMI≥30 AND at least one of the following:
   * Current/Previous smoking history ≥30 pack year
   * Chronic Obstructive Pulmonary Disease (COPD)
5. Female of childbearing potential should have a negative serum pregnancy test prior to index procedure.

   Note: All female of childbearing potential must agree to use a highly effective method of contraception (such as double barrier, oral or parenteral hormonal, intrauterine device and spermicide) consistently and correctly for the duration of the study.
6. Subject is willing and able to provide a signed Informed Consent Form and is willing and able to comply with study's procedures including follow-up visits.

Exclusion Criteria:

1. Subjects undergoing partial sternotomy.
2. Subjects with any preoperative active significant infection.
3. Subjects that received oral or IV doxycycline during the last 4 weeks prior to screening.
4. Subjects with sensitivity to doxycycline and/or to tetracycline family of drugs and/or other study drug ingredients.
5. Subjects with known allergies to more than 3 substances. (An allergy questionnaire will be filled during the screening process).
6. Subjects with history of allergic/hypersensitivity reaction to any substance having required hospitalization and/or treatment with intra-venous steroids/epinephrine or in the opinion of the investigator the patient is at high risk of developing severe allergic/hypersensitivity reactions.
7. Subjects with uncontrolled Asthma (GINA III-IV).
8. Subjects with chronic urticaria.
9. Immunocompromised subjects from any reason, at screening.
10. Subjects with renal failure requiring dialysis.
11. Subjects scheduled to major organ transplantation and/or to other significant concomitant surgical procedure.
12. Subjects scheduled for mechanical assist device.
13. Subjects scheduled to be treated with preventive negative pressure devices.
14. Subjects undergone Cerebro-Vascular Accident (CVA)/Transient Ischemic Attack (TIA) within the past 3 months prior to randomization.
15. Subjects that have undergone previously, any cardiac surgery through sternotomy.
16. Subjects with active or previous malignancy in the chest area.
17. Any subject with active malignancy or with malignancy that has not been in complete remission for at least 5 years. Subjects who have had carcinoma in situ of the cervix, squamous cell carcinoma of the skin and basal cell carcinoma of the skin, are eligible.
18. Pregnant or breast-feeding women or women of childbearing age not protected by an effective contraceptive method of birth control (such as double barrier, oral or parenteral hormonal, intrauterine device and spermicide).
19. Subjects enrolled in any intervention study with an investigational medicinal product and/or received any investigational medicinal product within 30 days or 5½ half-lives of the product prior to enrollment (whichever is longer).
20. In the opinion of investigator, subject is not eligible to participate in the study and/or to comply with protocol requirements (e.g. due to a cognitive, medical condition or residency distanced from site that may jeopardize Follow-Up visits attendance etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Sternal Wound Infection rate | within 90 days (3 months) post sternotomy for cardiac surgery
  Infection rate as measured by the proportion of subjects with a sternal wound infection event.
  Sternal wound infection is composed of Deep Sternal Wound Infection (DSWI) & Superficial Sternal Wound Infection (SSWI).
  Mortality from any reason within 90 days (3 months) post sternotomy, will be analyzed as treatment failure.

SECONDARY OUTCOMES:
Hospitalization days | 90 days
  Average number of Hospitalization days post sternotomy due to sternal infection.
Average ASEPSIS assessment score | 90 days (3 months) post sternotomy
  ASEPSIS (Additional treatment, Serous discharge, Erythema, Purulent exudate, Separation of deep tissue, Isolation of bacteria, Stay duration as inpatient), for wound assessment and treatment parameters, which provides numerically score during an inspection of the surgical site.
  The final score is being interpreted to severity of wound appearance and the clinical consequences of infections.
Number of surgical re-interventions | 90 days (3 months) post sternotomy
  Number of surgical re-intervention due to sternal surgical site infection.
Superficial Sternal Wound Infections (SSWI) | 90 days (3 months) post sternotomy
  Incidence of Superficial Sternal Wound Infections (SSWI)
Deep Sternal Wound Infections (DSWI) | 90 days (3 months) post sternotomy
  Incidence of Deep Sternal Wound Infections (DSWI)
Mortality rate associated with Sternal Wound Infection (SWI) | 90 days (3 months) post sternotomy
  Mortality rate associated with Sternal Wound Infection (SWI)
Determination of susceptibility to Doxycycline | 90 days (3 months) post sternotomy
  Determination of susceptibility to Doxycycline of any organism recovered from a Sternal Surgical Site Infection.

OTHER OUTCOMES:
Overall hospitalization days | 6 months
  Overall Hospitalization days, for any reason.
Readmission due to Sternal Surgical Site Infection | 90 days (3 months) post sternotomy
  Number of readmissions due to Sternal Surgical Site Infection
Time to Sternal Wound Infection | 90 days (3 months) post sternotomy
  Time to sternal wound infection (Post Operating Day) post sternotomy.
Analgesic treatment | 6 months
  Average number of analgesic treatment days
Visual Analogue Score (VAS) assessment | 6 months
  VAS score assessment, self-completed by the respondent, from 0 (no pain) to 10 (worst imaginable pain)
Antibiotic treatment due to Sternal Surgical Site Infections (all routes of administration). | 90 days (3 months) post sternotomy
  Average number of Antibiotic Treatment (overall IV and other administration modes, e.g. oral) days due to sternal Surgical Site Infection (SSWI & DSWI)
Antibiotic treatment due to Sternal Surgical Site Infections (IV administration). | 90 days (3 months) post sternotomy
  Average number of Antibiotic Treatment (IV administration) days due to sternal Surgical Site Infection (SSWI & DSWI)

CONTACTS AND LOCATIONS:
Overall Officials: Hartzell V. Schaff, M.D., Principal Investigator — Mayo Clinic, 220 First Street SW, Rochester, MN. 55902
Locations (3):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Hermann, Houston, Texas
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No